CLINICAL TRIAL: NCT00593021
Title: Diagnostic Evaluation of Obscure Gastrointestinal Bleeding
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, John Robinson Saltzman, MD, Director of Endoscopy, Brigham and Women's Hospital
Other Study IDs: SALTZMAN: 2007P-000991
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Obscure Gastrointestinal Bleeding
Keywords: Obscure Gastrointestinal Bleeding; Occult Gastrointestinal Bleeding; Overt Gastrointestinal Bleeding; Capsule Endoscopy; CT Enterography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Up to 5% of patients with recurrent gastrointestinal (GI) bleeding remain undiagnosed by EGD and colonoscopy, the presumed source of bleeding in these patients being the small intestine. These patients fall under the category of "obscure gastrointestinal bleeding," and frequently require an extensive diagnostic work-up. For these reasons, most patients who present with obscure or occult gastrointestinal bleeding typically undergo multiple endoscopic evaluations, including capsule endoscopy and various radiologic imaging studies, including enteroclysis, small bowel series, CT scan, angiography, and radionuclide scan. Recently, many centers (included the Brigham and Women's Hospital) have begun using capsule endoscopy and CT enterography (CTE) for evaluation of suspected small bowel pathology. This is an observational study enrolling patients referred to the Brigham and Women's Hospital for obscure gastrointestinal bleeding designed to compare the diagnostic yield of various diagnostic modalities, in particular capsule endoscopy and CT enterography in the evaluation of obscure gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Anemia, hematochezia, melena, Hematemesis, heme positive stool with negative EGD+/-colonoscopy

Exclusion Criteria:

* Under the age of 18
* Unable to give consent
* IV Contrast Allergy (excluded from CT)
* Renal insufficiency (excluded from CT)
* Unable to swallow (excluded from capsule)
* Small bowel obstruction or stricturing disease (excluded from capsule)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 and able to give consent who are referred to the Brigham and Women's Hospital Endoscopy Center or GI Clinic for the evaluation of obscure gastrointestinal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of capsule endoscopy and CT Enterography in patients with obscure GI bleeding | Continuous

SECONDARY OUTCOMES:
Hospital course, clinical improvement | 120 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: John R Saltzman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States